CLINICAL TRIAL: NCT01901198
Title: A Phase 1 Study to Evaluate the Pharmacokinetic and Pharmacodynamic Profile, Safety, and Tolerability of Escalating Single Dose Recombinant Human Serum Albumin/Interferon alpha2a Fusion Protein in Healthy Volunteers
Brief Title: Recombinant Human Serum Albumin/Interferon alpha2a Fusion Protein Phase I Study in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Bio-Fortune Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 921301
Record Dates: First submitted 2013-04-09; First posted 2013-07-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Serum Albumin, Human; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Human Serum Albumin/interferon alpha2a (Experimental): Human Serum Albumin/interferon alpha2a 300-1200 mcg single dose S.C.
  Interventions: Biological: Human Serum Albumin/interferon alpha2a 300-1200 mcg single dose S.C.
- Pegasys (Active Comparator): Peginterferon 180 mcg single dose S.C.
  Interventions: Biological: Peginterferon 180 mcg single dose S.C.

INTERVENTIONS:
Biological: Human Serum Albumin/interferon alpha2a 300-1200 mcg single dose S.C. — Recombinant Human Serum Albumin/interferon alpha2a Fusion Protein 300-1200 mcg at Day 0
  Arms: Human Serum Albumin/interferon alpha2a
Biological: Peginterferon 180 mcg single dose S.C. — Pegasys 180 mcg S.C. single dose on Day 0
  Arms: Pegasys

SUMMARY:
This study will evaluate safety, tolerability, pharmacokinetics and pharmacodynamics of Recombinant Human Serum Albumin/interferon alpha2a Fusion Protein single dose in Chinese healthy volunteers.

DETAILED DESCRIPTION:
This is an open-label study that will be conducted at a single site in China to characterize the PK/PD profile, safety and tolerability of Recombinant Human Serum Albumin/interferon alpha2a Fusion Protein in healthy subjects. Subjects will receive a single dose of Recombinant Human Serum Albumin/interferon alpha2a Fusion Protein or active comparator Pegasys at Day 0. The total duration of study participation is up to 6 weeks for each subject. Subjects will complete a follow-up visit at Day 28 after the dosing.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy males or females between 18 to 45 years old, inclusive
* Must have a body mass index (BMI) of 19 to 25 kg/m2, inclusive, and a minimum body weight of 50.0 kg

Exclusion Criteria:

* History of any clinically significant laboratory abnormalities, cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major diseases
* Female subjects who are pregnant or breastfeeding
* Any previous treatment with Human Albumin Interferon fusion protein

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events after single dose | 4 weeks

SECONDARY OUTCOMES:
Plasma concentration of interferon after single dose | 4 weeks
Plasma concentration of Neopterin after single dose | 4 weks

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, MD, Principal Investigator — Beijing YouAn Hospital
Locations (1):
- Beijing YouAn Hospital, Capital Medical University, Beijing, Beijing Municipality, China